CLINICAL TRIAL: NCT03175796
Title: Infant Mental Health-Home Visiting Randomized Controlled Trial
Acronym: IMH-HV RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Michigan Department of Health and Human Services (Other)
Responsible Party: Principal Investigator, Kate Rosenblum, Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM00124224
Record Dates: First submitted 2017-05-17; First posted 2017-06-05 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2021-11

CONDITIONS: Infant Mental Health

STUDY DESIGN:
Intervention Model Description: IMH-HV is a relationship-focused mental health intervention that aims to improve caregiver and child outcomes, including: improved caregiver mental health; enhanced positive parenting; decreased risk for physical/emotional neglect and/or abuse; and reduced risk for negative child outcomes including impaired development, cognitive delay and behavioral problems. In addition, IMH-HV services aim to reduce the probability of intergenerational transmission of the effects of unresolved loss and trauma in parents.
  The IMH-HV Model uses a range of strategies for intervention, such as:
  * attending to the health and basic material needs of the infant/toddler, parent(s), and family members;
  * providing developmental guidance for positive parenting behavior;
  * providing counseling/emotional support for the parents;
  * developing parents' life coping skills and social support; and
  * providing infant/parent psychotherapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IMH-HV Treatment Group (Experimental): Infant Mental Health-Home Visiting. Weekly home visits for up to one year by a trained IMH-HV treatment provider. Treatment delivery consistent with the IMH-HV manual.
  Interventions: Behavioral: Infant Mental Health-Home Visiting
- Treatment as Usual Control Group (No Intervention): No intervention provided as part of participation in this study; families are free to access community resources including any available treatment(s) in the community.

INTERVENTIONS:
Behavioral: Infant Mental Health-Home Visiting — Behavioral intervention aimed to increase parental competencies and promote mental health and sensitive caregiving.
  Arms: IMH-HV Treatment Group

SUMMARY:
The primary objective is to rigorously evaluate the effectiveness of the Infant Mental Health Home Visiting (IMH-HV) model on maternal and child outcomes according to legislative standards via a randomized controlled trial. The research team will recruit caregivers and their children (0-24 months) or pregnant women (n=72) from locations across Washtenaw County to participate in the IMH-HV RCT. Half of the women will be randomly assigned to a treatment as usual (TAU) control group (with access to all available community resources), and half of the women will be randomly assigned to the treatment group (i.e., IMH-HV). Women assigned to the control group will not receive IMH-HV treatment through the study team, but will not be prohibited from seeking or accessing IMH-HV treatment or any other services through community resources. Women assigned to the treatment group will receive IMH-HV treatment for 12 months through the study team with rigorous monitoring of fidelity to the IMH-HV model. All study participants will undergo assessments across the 24-month period (12 months of which are the treatment trial) (i.e., baseline (randomization will occur after baseline), mid-points (3, 6 and 9 months) and follow-ups (12, 18 and 24 months) after randomization). Additionally, all study participants will have the opportunity to participate in assessments regarding their experience of the COVID-19 pandemic.

The purpose of this study is to evaluate efficacy of the Infant Mental Health Home-Visiting (IMH-HV) model on parental and child outcomes according to legislative standards and consistent with the State of Michigan's benchmarks. If this study confirms the efficacy of the IMH-HV model, this will support the sustainability of IMH-HV in the state of Michigan as evidence from a randomized controlled trial is necessary in order to access certain state and federal dollars. Access to evidence-based and sustainable parenting support can ultimately improve outcomes for this vulnerable population. Specifically this study aims to:

1. Conduct a randomized controlled trial to evaluate the efficacy of IMH-HV treatment utilizing rigorous outcomes monitoring and evaluation methodology to establish that the families served achieve the intended positive benefit. Eligible caregivers and children or pregnant women will be assigned to the control group or the treatment group and both groups will receive research assessments at regular intervals measuring key impacts of the IMH-HV model.
2. Determine IMH-HV efficacy via analysis of treatment impact on key caregiver, child, and family indicators. The hypothesis is that there will be positive impacts of IMH-HV, with caregiver, child, and family-level improvements from baseline to post assessment on key indicators, including:

   1. Improved child outcomes as reflected in strengthened child physical and behavioral health, development and school readiness, and reduced risk for child maltreatment.
   2. Improved parental outcomes including improved parent mental health, decreased child abuse potential, and enhanced positive parenting.
   3. Improved family environment including decrease in crime and family violence, enhance linkage to referrals and improve family economics and self-sufficiency.
3. Identify factors associated with family improvement, including dosage and fidelity of treatment. It is the hypothesis that a dose-response association between the number of home visiting sessions and treatment impact, and a positive association between fidelity of treatment delivered and positive child and family outcomes.

DETAILED DESCRIPTION:
A small number of inclusion/exclusion criteria have not been disclosed in this record to preserve scientific integrity. They will be added to make this record complete once all study data is collected.

ELIGIBILITY:
Inclusion Criteria:

Mothers (biological or adoptive) who:

* are the permanent, primary caregiver of a child between the ages of 0-24 months old or 29+ weeks pregnant;
* are at least 18 years of age;
* who speak and understand English; and,
* who meet specified criteria for: childhood experiences, depression, challenges with child, and socio-economic status.

Exclusion Criteria:

* Women who live farther than 20 miles away from Ann Arbor
* Women who are already enrolled in Infant Mental Health-Home Visiting services
* Women who meet criteria for alcohol/substance use disorders, or who screen positive for psychosis

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Mothers that are primary, permanent caregivers of a child 0-24 months (male or female) OR 29+ weeks pregnant
Enrollment: 148 (Actual)
Dates: Start 2017-10-12 (Actual); Primary Completion 2020-08-17 (Actual); Study Completion 2020-08-17 (Actual)

PRIMARY OUTCOMES:
PTSD Checklist (PCL-5) | 1 Year
  Change in caregiver PTSD symptoms via measurement on PCL-5 with a range of 0 (no symptoms) to 80 (high level symptom endorsement).
Generalized Anxiety Disorder (GAD-7) | 1 Year
  Change in caregiver anxiety via measurement on GAD-7 with a range of 0 (no symptoms) to 21 (high level of anxiety symptoms endorsed).
Patient Health Questionnaire (PHQ-9) | 2 years
  Change in caregiver self-reported depression via measurement on PHQ-9 with a range of 0 (no depression symptoms) to 27 (high level of depression symptoms endorsed).
Brief Child Abuse Potential Inventory (BCAP) | 1 Year
  Change in caregiver self-reported emotional distress, rigidity, social isolation (risks associated with child maltreatment) via measurement on BCAP with a range of 0-24.
Working Model of the Child Interview (WMCI) | 1 year
  Categorization of caregiver perception of child and relationship with child that moves from distorted or disengaged to balanced via measurement on the WMCI.
Infant Toddler Social-Emotional Assessment (ITSEA) | 1 Year
  Change in caregiver reported social-emotional behavior problems of child via measurement on ITSEA using t-scores derived from ITSEA-provided standard norms

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Rosenblum, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Jester JM, Stacks AM, Riggs JL, Brophy-Herb HE, Muzik M, Rosenblum K; Michigan Collaborative for Infant Mental Health Research. Improved mental health for women receiving infant mental health home visiting: a randomized controlled trial. Front Psychol. 2025 Oct 9;16:1597655. doi: 10.3389/fpsyg.2025.1597655. eCollection 2025. PMID 41143010
- [Derived] Jones KA, Freijah I, Brennan SE, McKenzie JE, Bright TM, Fiolet R, Kamitsis I, Reid C, Davis E, Andrews S, Muzik M, Segal L, Herrman H, Chamberlain C. Interventions from pregnancy to two years after birth for parents experiencing complex post-traumatic stress disorder and/or with childhood experience of maltreatment. Cochrane Database Syst Rev. 2023 May 4;5(5):CD014874. doi: 10.1002/14651858.CD014874.pub2. PMID 37146219
- [Derived] Riggs JL, Rosenblum KL, Muzik M, Jester J, Freeman S, Huth-Bocks A, Waddell R, Alfafara E, Miller A, Lawler J, Erickson N, Weatherston D, Shah P, Brophy-Herb H; Michigan Collaborative for Infant Mental Health Research. Infant Mental Health Home Visiting Mitigates Impact of Maternal Adverse Childhood Experiences on Toddler Language Competence: A Randomized Controlled Trial. J Dev Behav Pediatr. 2022 May 1;43(4):e227-e236. doi: 10.1097/DBP.0000000000001020. Epub 2021 Oct 25. PMID 34698704